CLINICAL TRIAL: NCT03785041
Title: Comparative Study Between Preemptive and Postoperative Intra-articualr Injection of Levobupivacaine and Tramadol
Brief Title: Preemptive and Postoperative Intra-articualr Injection of Levobupivacaine and Tramadol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ayman Anis Metry, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASUH7923/16
Record Dates: First submitted 2018-12-19; First posted 2018-12-24 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Pain After Knee Arthroscop
Keywords: Tramadol; Intra-articular injection; Preemptive; post-arthroscopy pain; Levobupivacaine
MeSH Terms: interventions — Levobupivacaine; Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Levobupivacaine and tramadol Preemptive (Active Comparator): 20 ml 0.5% Levobupivacaine + 100 mg tramadol injected intraarticular preemptive.
  Interventions: Drug: Levobupivacaine Hydrochloride 2.5 MG/ML
- Tramadol and levobupivacaine postoperative (Active Comparator): 20 ml 0.5% Levobupivacaine + 100 mg tramadol injected intraarticular postoperative.
  Interventions: Drug: Levobupivacaine Hydrochloride 2.5 MG/ML
- Tramadol and levobupivacaine preemptive and postoperative (Active Comparator): 20 ml 0.25% Levobupivacaine + 50 mg tramadol injected intraarticular preemptive and postoperative.
  Interventions: Drug: Levobupivacaine Hydrochloride 2.5 MG/ML
- Levobupivacaine (Active Comparator): 20 ml 0.5% Levobupivacaine only injected intraarticular preemptive.
  Interventions: Drug: Levobupivacaine Hydrochloride 2.5 MG/ML

INTERVENTIONS:
Drug: Levobupivacaine Hydrochloride 2.5 MG/ML — Intrarticular injection of tramadol in addition to levobupivacaine in different doses preemptive and postoperative
  Other Names: Tramadol 50 MG/ML; Tramadol 100 MG/ML; Levobupivacaine Hydrochloride 5MG/ML

SUMMARY:
Comparison between preemptive and postoperative intraarticular injection of tramadol on pain sensation after arthroscopy

DETAILED DESCRIPTION:
220 patients assigned for therapeutic knee arthroscopy were divided into four equal groups in this prospective comparative study. All patients received IAI of 20 ml (0.5%) levopubivacaine alone in Group C; with 100 mg tramadol as PE (Group PE), at end of surgery (Group PO) or divided as 50 mg tramadol + 20 ml 0.25 % levobupivacaine as PE and 50 mg trmadol + 20 ml 0.25 % levobupivacaine as PO (Group PE/PO). Numeric rating scale (NRS) was used to assess pain sensation. Duration till request of rescue analgesia and number of requests were recorded. Patients' satisfaction concerning efficacy of PO analgesia was assessed using Iowa Satisfaction with Anesthesia Scale.

ELIGIBILITY:
Inclusion Criteria:

* Patient physical status according to American Society of Anesthesiology (ASA) classes I-II
* Patients free of general diseases prohibiting the use of local anesthesia.

Exclusion Criteria:

* Patients had allergy for local anesthetics or to tramadol
* Patients have psychological or neurological disorders inducing difficulty for evaluation of pain scoring.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Pain control | Pain assessment for 12 hours postoperative
  Pain sensation after arthroscopy assessed by numeric rating scale depending upon patient facial appearance with severe patient expressing high score and no pain with lowest score

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No